CLINICAL TRIAL: NCT07254780
Title: Effects of a Treatment Program Based on the Bobath Concept After Hospital Discharge in Children Born Very Preterm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, María del Mar Sánchez Joya, Phd Doctor, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BOBprem
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Premature Baby 26 to 32 Weeks; Premature Babies; Neurodevelopment Treatment; Neurodevelopment; Motor Disorder
Keywords: Physical Stimulation; Premature infant; Neurodevelopment; Neurodevelopment Treatment
MeSH Terms: conditions — Premature Birth; Motor Disorders | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TreatBOB (Experimental)
  Interventions: Other: Bobath
- TreatNO-BOB (Experimental)
  Interventions: Other: Early Intervention
- NoTreat-NO-BOB (Experimental)
  Interventions: Other: Ordinary care

INTERVENTIONS:
Other: Bobath — This group will receive an intervention based on the Bobath Concept, following the Bobath Clinical Reasoning Framework (BCRF). This approach adopts a holistic, systems-science perspective, considering the dynamic interaction between body functions, activities, participation, and contextual factors according to the ICF model.
  Arms: TreatBOB
Other: Early Intervention — This group will receive standard pediatric physiotherapy commonly implemented in early intervention services for children with motor disorders. The treatment will follow conventional approaches with a more impairment-based focus
  Arms: TreatNO-BOB
Other: Ordinary care — This group will receive ordinary care, defined as the standard protocol-based follow-up provided by the public health system, unrelated to Early Intervention physiotherapy services
  Arms: NoTreat-NO-BOB

SUMMARY:
INTRODUCTION: This project is presented as a continuation of the one approved in 2019 (Code: UALBIO2019/013). Early Intervention is defined as all interventions, including prevention, carried out with children aged 0-6 years, their families, and their environment, in order to respond to what each child needs to advance in their development as early as possible.

Psychomotor Delay indicates a slow developmental trajectory in several areas. Premature infants frequently face a potential psychomotor delay, usually due to the immaturity associated with being born earlier than expected. Children born preterm account for 50% of functional diversity in the pediatric population, presenting sequelae in the perinatal period, in the short term, and in the long term. In a previous study conducted by our group, the importance of early follow-up and treatment for children born very preterm was demonstrated.

Neurodevelopmental disorders with motor impairments in children require physiotherapy treatment from the time of diagnosis, throughout early childhood intervention, and across the lifespan. The most prevalent condition is cerebral palsy, which is the leading cause of childhood disability. Its prevalence ranges from 1.5 to 3.0 per 1,000 live births, with no major changes observed in adolescent and adult populations, and with higher occurrence in males than females. Other important conditions due to their frequency and symptoms include congenital malformations and syndromes.

OBJECTIVE: To analyze the effects of advanced physiotherapy programs on development, activity, and participation in children receiving early intervention and presenting motor disorders.

METHODOLOGY: Clinical trial with experimental groups and one control group. Advanced physiotherapy programs based on evidence will be studied, carried out with and involving the family, and supported by specialized care.

The sample will be obtained from centers and associations collaborating with the University of Almería. Before conducting the study, informed consent will be requested from parents or legal guardians. Baseline assessments and follow-up measurements will be performed. Validated and relevant variables related to development and motor difficulties will be used. The data obtained during the project will be stored in a database.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants with a gestational age between 24 and 32 weeks, with an adequate weight for their gestational age

Exclusion Criteria:

* Neurological disorders
* Invasive mechanical ventilation
* Congenital disorders
* Necrotising enterocolitis
* Metabolic diseases
* Intraventricular hemorrhage grade 3-4
* Genetic disorders
* Oral disorders that make this process difficult(cleft palate, cleft lip...)
* Serious illnesses according to medical criteria

Ages: 24 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-07-22 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
Gross Motor Skills | 2 Years
  To evaluate the baby's gross motor competence during early motor development, the investigators will employ the Alberta Infant Motor Scale (AIMS). This tool, developed by Canadian researchers, is an observational assessment designed for infants from birth until they achieve independent walking. It includes 58 items that examine antigravity muscle control and overall motor performance across four positions: prone, supine, sitting, and standing (de Albuquerque et al., 2015).
  This tool provides percentile scores (0-100) for gross motor developmental, with higher scores indicating more advanced abilities.
Neuromotor Development | 2 Years
  To evaluate motor, cognitive, and language development, the investigators will use the Bayley Scales of Infant and Toddler Development, Third Edition (Bayley-III), one of the most widely applied instruments for assessing early development. Its primary purpose is to identify children who may present developmental delays and to guide the planning of appropriate interventions. The Bayley-III consists of six subscales that measure cognitive, language, motor, social-emotional, adaptive, and behavioral skills in children aged 1 to 42 months (de Albuquerque et al., 2018).
  This tool provides percentile scores (0-100) for each developmental domain, with higher scores indicating more advanced abilities.

SECONDARY OUTCOMES:
Parents Experiences about Development | 2 Years
  To screen overall developmental progress, the investigators will use the Ages & Stages Questionnaires, Third Edition (ASQ-3). This parent-completed tool assesses children from 1 to 66 months across five domains: communication, gross motor, fine motor, problem-solving, and personal-social skills. Each questionnaire includes age-specific items that allow caregivers to report their child's abilities through simple observations.
  The ASQ-3 helps identify children who may need monitoring or further evaluation, providing a practical and reliable measure of early developmental functioning.
  This tool provides scores (0-60) for each developmental domain, with higher scores indicating more advanced abilities.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Almería, Almería, Spain

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available from the corresponding author upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available for one year once the study is finished
Access Criteria: Reasonable request to reproduce the intervention performed on this study

REFERENCES:
- [Background] Bernabe-Zuniga JE, Rodriguez-Lucenilla MI, Alias-Castillo AJ, Rueda-Ruzafa L, Roman P, Del Mar Sanchez-Joya M. Early interventions with parental participation and their implications on the neurodevelopment of premature children: a systematic review and meta-analysis. Eur Child Adolesc Psychiatry. 2025 Mar;34(3):853-865. doi: 10.1007/s00787-024-02528-1. Epub 2024 Jul 19. PMID 39028424
- [Background] Alonso-Fernandez S, de Liria CRG, Lluch-Canut T, Poch-Pla L, Perapoch-Lopez J, Juve-Udina ME, Martinez-Momblan MA, Hurtado-Pardos B, Roldan-Merino JF. Psychometric properties of the oral feeding assessment in premature infants scale. Sci Rep. 2022 May 12;12(1):7836. doi: 10.1038/s41598-022-11521-0. PMID 35551222
- [Background] de Albuquerque PL, Lemos A, Guerra MQ, Eickmann SH. Accuracy of the Alberta Infant Motor Scale (AIMS) to detect developmental delay of gross motor skills in preterm infants: a systematic review. Dev Neurorehabil. 2015 Feb;18(1):15-21. doi: 10.3109/17518423.2014.955213. Epub 2014 Oct 3. PMID 25279804
- [Background] Albuquerque PL, Guerra MQF, Lima MC, Eickmann SH. Concurrent validity of the Alberta Infant Motor Scale to detect delayed gross motor development in preterm infants: A comparative study with the Bayley III. Dev Neurorehabil. 2018 Aug;21(6):408-414. doi: 10.1080/17518423.2017.1323974. Epub 2017 May 24. PMID 28537470
- [Background] Seesahai J, Luther M, Church PT, Maddalena P, Asztalos E, Rotter T, Banihani R. The assessment of general movements in term and late-preterm infants diagnosed with neonatal encephalopathy, as a predictive tool of cerebral palsy by 2 years of age-a scoping review. Syst Rev. 2021 Aug 12;10(1):226. doi: 10.1186/s13643-021-01765-8. PMID 34384482